CLINICAL TRIAL: NCT07396467
Title: Clinical Characteristics, Prognosis, and Immunotherapy Outcomes in Patients With Lung Cancer and Concomitant Pulmonary Fibrosis: An Observational Study Integrated With Single-Cell and Spatial Transcriptomics
Brief Title: Clinical Outcomes and Immunotherapy in Lung Cancer With Pulmonary Fibrosis
Acronym: IPF-LC-IO
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IPF-LC-001
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer and Idiopathic Pulmonary Fibrosis
Keywords: Lung cancer, Pulmonary fibrosis, Immune checkpoint inhibitors (ICI), Tumor microenvironment (TME), scRNA-seq
MeSH Terms: conditions — Lung Neoplasms; Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lung cancer: patients with lung cancer without lung fibrosis
  Interventions: Other: there is no intervention
- lung cancer with lung fibrosis
  Interventions: Other: there is no intervention

INTERVENTIONS:
Other: there is no intervention — there is no intervention

SUMMARY:
This retrospective observational study will evaluate immune checkpoint inhibitor (ICI)-related outcomes in lung cancer patients with concomitant pulmonary fibrosis/interstitial lung disease (ILD) and determine how fibrosis/ILD modifies immunotherapy effectiveness and safety. We will characterize the clinical, radiographic, pathological, and molecular features of lung cancer with ILD and examine their associations with ICI response and survival. A comparator cohort of lung cancer patients without radiographic ILD from the same institution and time period will be used to compare ICI effectiveness (e.g., response and survival outcomes) and pulmonary toxicity signals, including pneumonitis/acute ILD exacerbation. In a translational sub-study, archived lung tumor specimens will undergo single-cell and spatial transcriptomic profiling to identify fibrosis-associated tumor-microenvironment programs that may underlie differential immunotherapy outcomes.

DETAILED DESCRIPTION:
Lung cancer with concomitant pulmonary fibrosis/interstitial lung disease (ILD) represents a clinically challenging population in whom immune checkpoint inhibitor (ICI) treatment may be influenced by baseline lung vulnerability and a distinct tumor immune microenvironment. This single-center, retrospective observational cohort study is designed to evaluate how fibrosis/ILD status and related clinical features are associated with immunotherapy use, effectiveness, and safety.

We will identify patients with pathologically confirmed lung cancer and radiographic evidence of pulmonary fibrosis/ILD diagnosed and treated at Jiangsu Province Hospital (The First Affiliated Hospital of Nanjing Medical University). A comparator cohort of lung cancer patients without radiographic ILD from the same institution and time period will be assembled to enable direct comparisons of immunotherapy outcomes. The study will characterize baseline demographics, smoking history, comorbidities, pulmonary function and imaging features (when available), tumor histology and stage, relevant laboratory indices, and molecular testing results. These variables will be examined for associations with ICI exposure and outcomes.

The primary analyses will focus on immunotherapy-related endpoints, including real-world measures of ICI effectiveness (such as objective response and survival outcomes captured in routine care) and ILD-relevant safety outcomes, including immune-related pneumonitis and/or acute exacerbation of underlying ILD, treatment interruption or discontinuation, and other clinically significant pulmonary adverse events. Comparative analyses will evaluate whether patients with lung cancer and fibrosis/ILD experience different ICI effectiveness or higher pulmonary toxicity risk compared with patients without ILD, and will explore which clinical, radiographic, pathological, or molecular features within the ILD cohort are linked to better or worse immunotherapy outcomes.

To investigate potential mechanisms underlying differential immunotherapy response in fibrosis-associated lung cancer, a translational sub-study will analyze available archived lung tumor specimens (e.g., bronchoscopic biopsy, CT-guided biopsy, or surgical samples). Single-cell transcriptomics and spatial transcriptomics will be performed to compare tumors arising in a fibrotic lung environment with tumors from patients without ILD. These analyses will be used to identify fibrosis-associated cellular states, immune microenvironment composition, and signaling programs that may contribute to altered immunotherapy sensitivity or toxicity. Findings from the multi-omics analyses will be integrated with clinical outcome data to generate mechanistic hypotheses and potential biomarkers relevant to immunotherapy decision-making in lung cancer patients with pulmonary fibrosis/ILD.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed lung cancer.

Interstitial lung disease (ILD) identified on chest imaging (e.g., HRCT).

Diagnosed and treated at Jiangsu Provincial People's Hospital between January 2019 and September 2025.

Exclusion Criteria:

* The anatomical location of the lung cancer lesion does not overlap with the ILD-involved area.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective, single-center observational cohort study of patients with pathologically confirmed lung cancer and imaging-confirmed interstitial lung disease (ILD) diagnosed at Jiangsu Provincial People's Hospital between January 2019 and September 2025. Eligible cases will be identified from hospital information systems and clinical records. Clinical characteristics, laboratory results, imaging, pathology and molecular reports will be extracted from HIS/LIS/PACS databases. Available tumor tissue specimens (bronchoscopic biopsy, CT-guided lung biopsy, or surgically resected lung tissue) will be collected for spatial transcriptomics analysis. Patients whose tumor location does not overlap with ILD-involved areas will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 24 months

SECONDARY OUTCOMES:
PFS | up to 24 months
ORR | up to 24 months

OTHER OUTCOMES:
AE | up to 24 months
  adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Nanjing medical university, Nanjing, China

IPD SHARING:
Plan to Share IPD: No